CLINICAL TRIAL: NCT03400202
Title: Eye Dark Circles: Physiopathologic Aspects and Influence on Quality of Life in Subjects of Various Ethnicities and Fitzpatrick Skin Types Utilizing Non-invasive In Vivo Instrumentation and Validated Questionnaires
Brief Title: Physiopathologic Aspects and Quality of Life in Participants With Eye Dark Circles
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRIC17-PHYEYE-01
Record Dates: First submitted 2018-01-11; First posted 2018-01-17 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Periorbital Hyperpigmentation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Group A: Dark Circles None: Group A includes participants with Dark Circle Severity Scale score 0 (None). Assessments of the participant's eye dark circles will be made after facial cleansing, utilizing in vivo skin imaging and quality of life questionnaires.
  Interventions: Device: Skin imaging; Other: Facial cleanser
- Group B: Dark Circles Mild: Group B includes participants with Dark Circle Severity Scale score 1 to 3 (Mild). Assessments of the participant's eye dark circles will be made after facial cleansing, utilizing in vivo skin imaging and quality of life questionnaires.
  Interventions: Device: Skin imaging; Other: Facial cleanser
- Group C: Dark Circles Moderate: Group C includes participants with Dark Circle Severity Scale score 4 to 6 (Moderate). Assessments of the participant's eye dark circles will be made after facial cleansing, utilizing in vivo skin imaging and quality of life questionnaires.
  Interventions: Device: Skin imaging; Other: Facial cleanser
- Group D: Dark Circles Severe: Group D includes participants with Dark Circle Severity Scale score 7 to 9 (Severe). Assessments of the participant's eye dark circles will be made after facial cleansing, utilizing in vivo skin imaging and quality of life questionnaires.
  Interventions: Device: Skin imaging; Other: Facial cleanser

INTERVENTIONS:
Device: Skin imaging — Non-invasive in vivo skin imaging will be taken with the VivoSight Ox Optical Coherence Tomography (OCT).
Other: Facial cleanser — Facial cleanser prior to procedures.
  Other Names: SkinMedica Facial Cleanser

SUMMARY:
This study will evaluate the physiopathologic characteristics of dark circles in participants with various ethnicities and Fitzpatrick Skin Types and the impact of the dark circles on the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Fitzpatrick skin type I-VI
* Willingness to not wear any eye makeup on the day of the study visit prior to the study visit appointment
* Willingness to cleanse the face and remove all makeup at least 15 minutes prior to each scheduled clinic visit
* Willingness to have facial exams, skin instrumentation measurements, and digital photos performed on the face.

Exclusion Criteria:

* Individuals with active symptoms of allergy, cold sore or warts, active psoriasis or eczema, rosacea, sunburn, open wounds, neurotic excoriations, excessive scarring, tattoos, or other skin conditions in the test area
* Uncontrolled disease such as diabetes, hypertension, hyper or hypo-thyroidism, active hepatitis, immune deficiency, or autoimmune
* Individuals who have a pre-existing or dormant dermatologic condition (e.g. history of severe psoriasis, atopic dermatitis, rosacea, skin cancer, etc.)
* Individuals who have had a blepharoplasty procedure or any other surgery in proximity or affecting the test area
* Individuals with recent procedures/surgeries (less than 6 months) on the eye bulb
* Individuals with permanent makeup around the eye area
* Chemical peel, microdermabrasion, microneedling, or dermaplaning in the previous 4 weeks
* Latisse, Revitalash, or other lash enhancement stimulators in the previous 1 month
* Retin-A®, Retin-A Micro®, Renova®, Avita®, Tazorac®, Avage® or Differin® or other similar prescription drugs within the previous 3 months
* Cosmetic injections (filler and/or toxins, i.e.Juvederm, Radiesse, Botox, etc.), non- ablative laser or fractional laser resurfacing in the previous 12 months
* Accutane® or other oral retinoid, Ablative procedures (i.e. laser, chemical) in the previous 12 months
* Individuals who have any planned surgeries or procedures during the study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants at a Clinical Research Center.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Dark Circles Severity Scale Score | Day 1
  The investigator will access the participant's lower and upper eyelids using the Dark Circles Severity Scale where 0=None to 9=Severe (very dark circles).
Classification Type of Dark Circles Score | Day 1
  The investigator will assess the lower eyelids for the following types of dark circles: Pigmented, Vascular and Shadow Effect. Each of these 3 types are graded where 0=none to 3=severe.

SECONDARY OUTCOMES:
Subject Questionnaire on Dark Circles, Medical History, and Lifestyle Habits | Day 1
  The Subject Questionnaire on Dark Circles, Medical History and Lifestyle Habits is a 15-item questionnaire completed by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goberdhan, Study Chair — Allergan
Locations (1):
- SkinMedica Clinical Research and Innovation Center, Irvine, California, United States

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_AGN_7181&studyid=641&filename=20180209%20CT.gov%20PRF%20Update%20Receipt%20SCRIC17-PHYEYE-01.pdf